CLINICAL TRIAL: NCT03869801
Title: Comparison of Ultrasound Guided Bilateral Erector Spinae Plane Block and Quadratus Lumborum Block in Laparoscopic Cholecystectomy
Brief Title: Comparion of Erector Spinae Plane Block and Quadratus Lumborum Block in Laparoskopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Asst. Prof. Serkan Tulgar, M.D., associate professor in anesthesiology, Maltepe University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ESP vs QLB in LC
Record Dates: First submitted 2019-03-08; First posted 2019-03-11 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Postoperative Pain; Anesthesia, Local
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Block (Active Comparator)
  Interventions: Procedure: erector spinae plane block
- QLB block (Active Comparator)
  Interventions: Procedure: quadratus lumborum block

INTERVENTIONS:
Procedure: erector spinae plane block — Ultrasound-guided bilateral Erector spinae plane (ESP) block performed before the surgery. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Other Names: Standard Pain Followup and Monitorization
  Arms: ESP Block
Procedure: quadratus lumborum block — Ultrasound-guided bilateral Quadratus lumborum (QLB) type 2 block performed before the surgery. Perioperative and postoperative routine analgesic protocol will be performed (consist of intravenous analgesics and intravenous patient-controlled analgesia) with no additional intervention (block) Standard Pain Followup and Monitorization will be performed.
  Other Names: Standard Pain Followup and Monitorization
  Arms: QLB block

SUMMARY:
Erector Spinae Plane Block is a newly defined regional anesthesia technique. Its use for many indications has been identified by case reports in the literature. As the investigators have considered that erector spinae plane block could be efficacious for providing postoperative analgesia in laparoscopic cholecystectomy, the investigators have implemented the application of this blockade into practice at the clinic.Quadratus Lumborum block (QLB) type 2 is another regional anesthesia technic used for postoperative analgesia in laparoscopic cholecystectomy. Main purpose of this study is to compare the analgesic effect of ultrasound-guided erector spinae block and QLB in laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Elective laparoscopic Cholecystectomy, ASA status 1-2

Exclusion Criteria:

* Patient refusal Contraindications to regional anesthesia Known allergy to local anesthetics Bleeding diathesis Use of any anti-coagulants Inability to provide informed consent Severe kidney or liver disease Inability to operate PCA system Patient with psychiatric disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
analgesic consumption | 24 hours
  opioid consumption in Patient Controlled Analgesia device

SECONDARY OUTCOMES:
NRS scores | 24 hours
  Changes in Numeric Rating Scale (NRS) at rest and on movement will be recorded at intervals. NRS is a unidimensional measure of pain intensity in adults. The NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").

CONTACTS AND LOCATIONS:
Locations (3):
- Turkey (Türkiye) (3):
  - Antalya research hospital, Antalya
  - Maltepe University faculty of medicine, Istanbul
  - Cigli Educatinal Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okmen K, Metin Okmen B, Topal S. Ultrasound-guided posterior quadratus lumborum block for postoperative pain after laparoscopic cholecystectomy: A randomized controlled double blind study. J Clin Anesth. 2018 Sep;49:112-117. doi: 10.1016/j.jclinane.2018.06.027. Epub 2018 Jun 18. PMID 29929169
- [Result] Tulgar S, Kapakli MS, Senturk O, Selvi O, Serifsoy TE, Ozer Z. Evaluation of ultrasound-guided erector spinae plane block for postoperative analgesia in laparoscopic cholecystectomy: A prospective, randomized, controlled clinical trial. J Clin Anesth. 2018 Sep;49:101-106. doi: 10.1016/j.jclinane.2018.06.019. Epub 2018 Jun 15. PMID 29913392